CLINICAL TRIAL: NCT05625607
Title: Evaluation of Clinical Outcomes of Transcatheter Transfemoral Mitral Valve-in-Valve Implantation in Polish Population- Observational Multicenter Registry
Brief Title: Polish Transcatheter Transfemoral Mitral Valve-in-Valve Implantation (Mitral ViV) Registry
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: National Institute of Cardiology, Warsaw, Poland (Other); Medical University of Bialystok (Other); University of Opole (Other); Medical University of Gdansk (Other); Medical University of Silesia (Other); Medical University of Lodz (Other)
Responsible Party: Sponsor
Other Study IDs: WUM-MViV
Record Dates: First submitted 2022-11-02; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Mitral Insufficiency; Mitral Stenosis; Mitral Stenosis With Insufficiency; Heart Failure; Bioprosthesis Failure
Keywords: Transcatheter mitral valve replacement; Transcatheter mitral valve implantation; Mitral valve-in-valve; Mitral valve insufficiency; Mitral stenosis; Mitral regurgitation; Bioprosthesis failure; Left ventricle outflow tract obstruction
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Procedure: Transcatheter mitral valve-in-valve implantation — Transcatheter transfemoral mitral valve-in-valve implantation is an alternative for surgery redo in high-surgical-risk patients with bioprosthetic valve failure. The procedure is performed via femoral vein access. By the transseptal puncture (in the postero-inferior part of the interatrial septum) and balloon septostomy, the bioprosthetic valve is introduced through the degenerative valve into the left ventricle. The valve is expanded in the mitral position during rapid ventricle pacing.

SUMMARY:
In recent years increasing number of mitral bioprosthesis implantation, especially in elderly population, is observed. Bioprosthetic valves are associated with a lower risk of thrombotic and bleeding adverse events compared with mechanical prostheses, but their use is limited due to their durability. After years numerous patients may develop bioprosthesis failure, requiring valve reintervention. Significantly burdened ones are oftentimes disqualified or not referred to surgery redo. An emerging treatment method for these patients is transcatheter mitral valve-in-valve implantation as an alternative to re-operation. This technique is applied with the use of devices previously dedicated to transcatheter aortic valve implantation (TAVI). Recent papers prove that transcatheter mitral valve replacement (TMVR) is a safe and effective procedure when performed in a selected group of high-surgical-risk patients. However, data regarding the Polish population are limited. Therefore, the aim of the study is to create a nationwide registry, collecting data from all Polish centers performing TMVR in order to describe the population of patients developing mitral bioprosthesis failure, evaluate their follow-up after TMVR as well as results of the transcatheter valvular intervention and identify potential limitations of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Failing surgically implanted mitral bioprosthetic valve demonstrating ≥ moderate stenosis and/or ≥ moderate insufficiency
* Qualification for TMVR by decision of the local Heart Team
* Patient provided written informed consent

Exclusion Criteria:

- Disqualification from TMVR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Polish patients with failed surgically implanted mitral bioprosthetic valves, qualified by decision of the Heart Team to TMVR. All patients meeting inclusion criteria will prospectively included in the study. Patients meeting inclusion criteria before the set-up of registry will be included retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality | 1 year
  Endpoint described as n=x (y%).
Rate of hospitalization | 1 year
  Hospitalization for valve-related symptoms or worsening congestive heart failure.
  Endpoint described as n=x (y%).
Rate of neurological events | 1 year
  All stroke, transient ischemic attack (TIA). Endpoint described as n=x (y%).
Rate of myocardial infarction | 1 year
  Endpoint described as n=x (y%).
Rate of valve-related dysfunction | 1 year
  Mean transvalvular gradient ≥5mmHg; ≥mitral regurgitation; ≥mild paravalvular leak; left ventricle outflow tract obstruction (LVOTO)- (acute hemodynamic deterioration associated with imaging evidence of LVOTO; mean LVOT pressure gradient increasement ≥10 mmHg compared to the baseline value).
  Endpoint described as n=x (y%).

SECONDARY OUTCOMES:
Rate of technical success | at 24 hours
  Absence of procedural mortality; successful access, delivery, and retrieval of the device delivery system; successful deployment and correct positioning of the first intended device; freedom from emergency surgery or reintervention related to the device or access procedure.
  Endpoint described as n=x (y%).
Rate of device success | 30 days, 6 month, 1 year
  Absence of procedural mortality or stroke; proper placement and positioning of the device; freedom from unplanned surgical or interventional procedures related to the device or access procedure; continued intended safety and performance of the device.
  Endpoint described as n=x (y%).
Rate of procedural success | 30 days
  Device success (either optimal or acceptable), and absence of major device or procedure related serious adverse events, including:
  A. Death B. Stroke C. Life-threatening bleeding (Mitral Valve Academic Research Consortium scale) D. Major vascular complications E. Major cardiac structural complications F. Stage 2 or 3 acute kidney injury (includes new dialysis) G. Myocardial infarction or coronary ischaemia requiring PCI or CABG H. Severe hypotension, heart failure, or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for ≥48 h.
  I. Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention Endpoint described as n=x (y%).
Rate of patient success | 1 year
  I. Device success; II. Patient returned to the pre-procedural setting; III. No rehospitalizations or reinterventions for the underlying condition; IV. Improvement from baseline in symptoms; improvement by ≥1 functional class in New York Heart Association scale. Nominal values from I to IV, where higher value indicates worse outcome; V. Improvement from baseline in functional status; improvement by ≥50 m in 6-min walk test. Continuous values in meters, where higher value indicates better outcome; VI. Improvement from baseline in quality-of-life; improvement by ≥10 in Kansas City Cardiomyopathy Questionnaire. Scores are scaled from 0 to 100, where higher value indicates better outcome.
  Endpoint described as n=x (y%).

CONTACTS AND LOCATIONS:
Locations (7):
- Poland (7):
  - Medical University of Białystok, Bialystok
  - Medical University of Gdańsk, Gdansk
  - Medical University of Silesia, Katowice
  - Medical University of Łódź, Lodz
  - Medical University of Opole, Opole
  - Medical University of Warsaw, Warsaw
  - Institute of Cardiology, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone GW, Adams DH, Abraham WT, Kappetein AP, Genereux P, Vranckx P, Mehran R, Kuck KH, Leon MB, Piazza N, Head SJ, Filippatos G, Vahanian AS; Mitral Valve Academic Research Consortium (MVARC). Clinical trial design principles and endpoint definitions for transcatheter mitral valve repair and replacement: part 2: endpoint definitions: A consensus document from the Mitral Valve Academic Research Consortium. Eur Heart J. 2015 Aug 1;36(29):1878-91. doi: 10.1093/eurheartj/ehv333. Epub 2015 Jul 13. PMID 26170468